CLINICAL TRIAL: NCT01758367
Title: Decitabine Followed by Donor Lymphocyte Infusion for Patients With Relapsed Acute Myeloblastic Leukemia(AML) After Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li Yu, Director of Department of Hematology, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN301-XYK-002
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia
Keywords: demethylating agent; immunogenicity; decitabine(DAC); donor lymphocyte infusion(DLI); AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

ARMS (1):
- Decitabine+DLI (Experimental): Patients with relapsed AML after Allo-HSCT will be treated with decitabine and DLI.
  Interventions: Drug: Deciatbine(DAC)

INTERVENTIONS:
Drug: Deciatbine(DAC)
  Other Names: 5-aza-2'-deoxycytidine

SUMMARY:
Decitabine can up-regulate a series of immune associated proteins, including cancer testis antigens (CTA), major histocompatibility complex (MHC), co-stimulatory molecules and adhesion molecules, which suggests a potential benefit for a following adoptive T cell therapy. In addition, decitabine induce FOXP3 expression in CD4+ T cells and convert CD4+ T cells into T regulatory cells(Tregs). As a result, Graft versus host disease(GVHD) can be reduced by treatment of decitabine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* Histologically or cytologically documented relapse of acute myeloid leukemia after a stem cell transplant
* Must have the ability to observe the efficacy and events
* Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Must have suitable donor

Exclusion Criteria:

* Must not have an advanced malignant hepatic tumor
* Must not receive any other forms of chemotherapy after cell infusion during the treatment protocol
* Must not be receiving any other investigational agents within 14 days of first dose of study drug
* Must not have uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Must not be pregnant or breastfeeding; pregnant women are excluded from this study because decitabine is a Category D agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine; these potential risks may also apply to other agents used in this study
* Must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or other agents used in the study
* Must not have a known or suspected hypersensitivity to decitabine
* Must not be human immunodeficiency virus (HIV)-positive and on combination antiretroviral therapy; these patients are ineligible because of the potential for pharmacokinetic interactions with decitabine; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 4 months

SECONDARY OUTCOMES:
overall survival | 3 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China